CLINICAL TRIAL: NCT07364058
Title: Assessment of Platelet-derived GARP in Atherosclerotic Disease
Acronym: CAPGAD
Status: Not yet recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Other Study IDs: CAPGAD
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atheroma; Carotid Artery; Atheromatosis
Keywords: Atheroma; Atherosclerosis; GARP; LRRC32
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis; Plaque, Atherosclerotic | interventions — Histocompatibility Testing; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The plaques extracted from carotid or femoral endarterectomy will be used or all analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endarterectomy population: This group includes patients with significant atherosclerotic burden justifying a surgical intervention of carotid or femoral endarterectomy.
  Interventions: Other: Tissue sample and data collection

INTERVENTIONS:
Other: Tissue sample and data collection — Tissue sample and data collection

SUMMARY:
The leading cause of death is cardiovascular diseases in occidental countries. Of those, atherosclerosis is the major contributor to this burden being notably responsible for strokes and myocardial infarctions. The genesis of atherosclerosis is linked to both lipid accumulation and inflammation in the vascular wall of major arteries. One of the major pathways of inflammation is the TGF-beta axis which is at least partially regulated by the GARP protein. It has been investigated mostly in cancer biology but data in cardiovascular disease is lacking. Thus, the investigators aim to characterize the contribution of this protein by investigating its expression in tissue from patients with atherosclerosis, the carotid or femoral plaque representing a good source of residual material adequate for research purpose. The main cells expressing the GARP protein are the platelets and the T regulating cells which will be the main focus.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Able to give informed consent
* Undergoing carotid or femoral endarterectomy

Exclusion Criteria:

* Younger than 18 years
* Pregnant
* Dialysis
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients undergoing femoral or carotid endarterectomy in our tertiary care center (Cliniques Universitaires Saint-Luc) for atherosclerotic disease who do not meet exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
GARP Expression in Platelets | Throughout the entire study, approximately during 3 years
  The number of cells/area expressing the GARP protein will be assessed

SECONDARY OUTCOMES:
GARP Expression T Regulating Cells | Throughout the entire study, approximately during 3 years
  The number of cells expressing GARP will be assessed as a number of cells / area
GARP Expression General | Throughout the entire study, approximately during 3 years
  The type of cells expressing GARP will be assessed as a number of cells / area

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Beauloye, Medical Degree, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No